CLINICAL TRIAL: NCT04707950
Title: Use of Tranexamic Acid for the Prevention of Postpartum Haemorrhage After Cesarean Section in High-risk Patients ( a Randomized Control Trial ).
Brief Title: Tranexamic Acid for the Prevention of Postpartum Haemorrhage
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Dr. Abou Bakr Mohamed El Nashaar, Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEAbdelfattah
Record Dates: First submitted 2020-02-25; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Postpartum Hemorrhage
Keywords: Tranexamic acid; postpartum hemorrhage; cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups: a study group & a control group. In addition to the standard management, the study group will be given TXA 1 gm (100 mg/ml) slowly intravenous infusion during delivery after clamping of the cord (administered over 10 minutes at 1 ml/minute).
  The second dose of TXA 1 g Intravenous can be given if:
  * Bleeding continues after 30 minutes
  * Bleeding restarts within 24 hours of completing the first dose While the control group will not be given TXA and we will compare the results in both groups (amount of blood loss during operation to assess the efficacy of TXA in the prevention of PPH and reduction of intraoperative and postoperative blood loss and to assess its safety and benefit in the reduction of incidence of hysterectomy or blood transfusion requirements).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group will be given tranexamic acid (Active Comparator): Participants will be divided into two groups: a study group & a control group. In addition to the standard management, the study group will be given TXA 1 gm (100 mg/ml) slowly intravenous infusion during delivery after clamping of the cord (administered over 10 minutes at 1 ml/minute).
  The second dose of TXA 1 g Intravenous can be given if:
  * Bleeding continues after 30 minutes
  * Bleeding restarts within 24 hours of completing the first dose While the control group will not be given TXA and we will compare the results in both groups (amount of blood loss during operation to assess the efficacy of TXA in the prevention of PPH and reduction of intraoperative and postoperative blood loss and to assess its safety and benefit in the reduction of incidence of hysterectomy or blood transfusion requirements).
  Interventions: Drug: Tranexamic Acid 100 milligram/Milliliter; Drug: Oxytocin
- Control group (Placebo Comparator): The control group will not be given Tranexamic acid but only the standard management ( Oxytocin )
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Tranexamic Acid 100 milligram/Milliliter — Participants will be divided into two groups: a study group & a control group. In addition to the standard management, the study group will be given TXA 1 gm (100 mg/ml) slowly intravenous infusion during delivery after clamping of the cord (administered over 10 minutes at 1 ml/minute).
  The second dose of TXA 1 g Intravenous can be given if:
  * Bleeding continues after 30 minutes
  * Bleeding restarts within 24 hours of completing the first dose While the control group will not be given TXA and we will compare the results in both groups (amount of blood loss during operation to assess the efficacy of TXA in the prevention of PPH and reduction of intraoperative and postoperative blood loss and to assess its safety and benefit in the reduction of incidence of hysterectomy or blood transfusion requirements).
  Other Names: Study group
  Arms: study group will be given tranexamic acid
Drug: Oxytocin — both groups will be given oxytocin as a standard management
  Other Names: Control group

SUMMARY:
Use of tranexamic acid (TXA) for the prevention of postpartum haemorrhage (PPH) after cesarean section in high-risk patients ( a randomized control trial ).

DETAILED DESCRIPTION:
Participants will be divided into two groups: a study group & a control group. In addition to the standard management, the study group will be given TXA 1 gm (100 mg/ml) slowly intravenous infusion during delivery after clamping of the cord (administered over 10 minutes at 1 ml/minute).

The second dose of TXA 1 g Intravenous can be given if:

* Bleeding continues after 30 minutes
* Bleeding restarts within 24 hours of completing the first dose While the control group will not be given TXA and we will compare the results in both groups (amount of blood loss during operation to assess efficacy of TXA in prevention of PPH and reduction of intra and postoperative blood loss and to assess its safety and benefit in the reduction of incidence of hysterectomy or blood transfusion requirements).

ELIGIBILITY:
Inclusion Criteria:

Scheduled or unscheduled cesarean delivery. Singleton or twin gestation.

Women at high risk for PPH after cesarean section:

Placenta previa, accreta, increta or percreta. haematocrit (HCT) < 30%. Bleeding at admission. History of Postpartum haemorrhage. Abnormal vital signs (hypotension or tachycardia). Previous Cesarean or uterine surgery. More than four previous deliveries. Multiple Gestation. Large Uterine fibroids. Chorioamnionitis. Magnesium sulphate use. Prolonged use of oxytocin.

Exclusion Criteria:

1. Age less than 18 years.
2. Women who are not at high risk for PPH.
3. Women attending for normal vaginal delivery.
4. Pre-existing maternal hemorrhagic conditions such as Factor 8 deficiency - haemophilia A carrier, Factor 9 deficiency - haemophilia B carrier or Von Willebrand's disease.
5. Recent diagnosis or history of venous thromboembolism or arterial thrombosis because TXA is a risk factor for thromboembolism, and its use is contraindicated.
6. Known congenital or acquired thrombophilias, including antiphospholipid antibody syndrome, because of the increased risk of thrombosis.
7. Autoimmune diseases such as lupus, rheumatoid arthritis, Sjogren's disease, and inflammatory bowel disease because of hypercoagulability and the increased risk of thrombosis or thromboembolism
8. Need for a therapeutic dose of anticoagulation before delivery, because the risk of thrombosis may be increased with TXA.
9. Hypersensitivity to TXA or any of its ingredients.
10. Transfusion or planned transfusion of any blood products during the current admission because the primary outcome is already pre-determined and the need for transfusion will be unrelated to perioperative haemorrhage
11. Seizure disorder (including eclampsia), and its use has been associated with postoperative seizures..
12. Active cancer, because of the risk of thromboembolism.
13. Congestive heart failure requiring treatment, because of the risk of thrombosis.
14. If there is no haemoglobin and hematocrit result available from the last 4 weeks since it is necessary to measure the postoperative change in haemoglobin and hematocrit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with high risk for postpsrtum hemorrhage after ceserean section
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-25 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Volume of blood loss | 30 minutes after baby delivery
  150 ml/pack

SECONDARY OUTCOMES:
transfusion requirements | 7 days postpartum
  number of women transfused blood
additional medical intervention | 48 hours postpartum
  number of patients were treated by an additional medical intervention
additional surgical or radiological interventions to control bleeding | 7 days postpartum
  number of patients were treated by additional surgical or radiological intervention
Change in maternal hematocrit concentration | 48 hours postpartum
  Hematocrit concentration (Percent)
Tranexamic acid side effects | 24 hours postpartum
  number of patients suffered from side effects
thromboembolic events | 7 days postpartum
  number of patients suffered from thromboembolic events
Maternal death | 7 days postpartum
  Number of women will die.

CONTACTS AND LOCATIONS:
Overall Officials: Abubaker M Elnashar, MD, Principal Investigator — Benha Faculty of Medecine
Locations (2):
- Egypt (2):
  - Benha university hospital, Banhā, Banha
  - Benha University, Banhā, Banha

IPD SHARING:
Plan to Share IPD: No